CLINICAL TRIAL: NCT04385186
Title: Inactivated Convalescent Plasma as a Therapeutic Alternative in Hospitalized Patients CoViD-19
Brief Title: Inactivated Convalescent Plasma as a Therapeutic Alternative in Patients CoViD-19
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Blood Center Foundation, Hemolife (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CT01
Record Dates: First submitted 2020-05-06; First posted 2020-05-12 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Infections, Coronavirus
Keywords: CoViD-19; Pathogen inactivation; Apheresis; Convalescent plasma
MeSH Terms: conditions — Coronavirus Infections; COVID-19 | interventions — Extracorporeal Membrane Oxygenation

STUDY DESIGN:
Intervention Model Description: MULTICENTER, CONTROLLED, RANDOMIZED, SIMPLE BLIND, CLINICAL TRIAL
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Convalescent plasma+Support treatment selected by the hospital (Experimental): Participants will receive two doses of ABO - Rh compatible inactivated convalescent plasma, each one of 200 mililiters (mL), with a 24-hour interval via transfusion, for a final volume of 400 mL, meanwhile they continue to receive the supportive treatment chosen by the hospitals, according to each institutional protocol.
  Interventions: Drug: Inactivated convalescent plasma; Drug: Support treatment
- Support treatment selected by the hospital (Active Comparator): The best support treatment selected by the hospital, according to each institutional protocol. Due to the ongoing development of knowledge of pathophysiology and scientific evidence of the available alternatives, it will be selected at the time of treatment.
  Interventions: Drug: Support treatment

INTERVENTIONS:
Drug: Inactivated convalescent plasma — Day 0: Transfusion of 200mL of ABO -Rh compatible inactivated convalescent plasma, Start of support treatment selected by medical staff according to each institutional protocol
  Day 1: Transfusion of 200mL of ABO -Rh compatible inactivated convalescent plasma
  Other Names: Inactivated convalescent plasma SARS-Cov-2 + Support treatment
  Arms: Convalescent plasma+Support treatment selected by the hospital
Drug: Support treatment — Day 0: Start of support treatment selected by medical staff according to each each institutional protocol
  Other Names: Support treatment under medical decision

SUMMARY:
Convalescent plasma is a way to provide passive immunity to a person exposed to an infectious agent. It has been used as a therapeutic tool for emerging viral infections without specific treatment and with high morbidity and mortality, such as Influenza H1N1, H5N1, H7N9, Ebola, MERS, SARS-CoV1, and even SARS-Cov2, with satisfactory results regarding evolution clinic of patients treated and without significant adverse events reported. One of its main advantages of convalescent plasma is to generate a rapid immune response (even faster than a vaccine), against a pathogen that circulates in a specific geographic area, probably common for both donor and recipient.

DETAILED DESCRIPTION:
This study consists of obtaining convalescent plasma by means of apheresis, from recovered donors, who meet the eligibility criteria to donate. Then this plasma will be inactivated by riboflavin and UV based photochemical treatment (Mirasol technology - Terumo BCT®), in order to add more transfusion security to the procedure. Finally, it will be transfused to CoViD-19 patients hospitalized in any of the participating clinics. There are currently no reported significant adverse events associated with this therapy. Have been published two serial cases reports,more evidence is necessary to standardize the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Confirmed laboratory diagnosis for qRT-PCR to SARS-CoV-2
* Meet any of the following medical criteria (Defined by WHO): Be currently hospitalized with: Pneumonia, Severe pneumonia, Acute Respiratory Distress Syndrome (moderate or severe), Sepsis or Septic shock
* The patient, or his representative, must sign an informed consent

Exclusion Criteria:

* Participate in another clinical trial for CoViD- 19
* History of acute allergic transfusion reactions due to transfusion of blood or other components, especially plasma components (fresh frozen plasma, cryoprecipitate and platelets),
* History of allergic reaction due to IgA deficiency
* Allergic reaction to sodium citrate or riboflavin (vitamin B2)
* History of immunosuppression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-06-20 (Estimated); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Mortality reduction in CoViD-19 patients treated with inactivated convalescent plasma + support treatment | Over a period of 28 days
  To assess the efficacy in reducing mortality in CoViD-19 patients treated with inactivated convalescent plasma together with the support treatment selected by the respective hospital

SECONDARY OUTCOMES:
Clinical evolution | Over a period of 28 days
  Number of Participants with resolution of fever (<38ºC temperature)
Clinical evolution by seven-parameter ordinal scale | 3, 7, 14 and 28 days
  The clinical improvement will be established with a two-point improvement within this seven categories (recommended by World Organization Health-WHO): 1) Not hospitalized, with resumption of normal activities 2) Not hospitalized, but unable to resume normal activities 3) Hospitalized that does not require supplemental oxygen 4) Hospitalized requiring supplemental oxygen 5) Hospitalized requiring high-flow nasal oxygen therapy, non-invasive mechanical ventilation, or both 6) Hospitalized requiring extracorporeal membrane oxygenation, invasive mechanical ventilation, or both 7) death
Multi-organ failure progression | 3, 7, 14 and 28 days
  Evolution by SOFA (Sequential Organ Failure Assessment), The range is between 0 and 24 points, with the highest scores being indicators of a more serious illness
Change in hemoglobin concentration | 3, 7, 14 and 28 days
  Compare the change in hemoglobin concentration at 3, 7, 14 and 28 days after treatment
Change in blood cell count | 3, 7, 14 and 28 days
  Compare the change in blood cell count at 3, 7, 14 and 28 days after treatment
Change in serum creatinine level | 3, 7, 14 and 28 days
  Compare the change in Serum creatinine concentration at 3, 7, 14 and 28 days after treatment
Change in aspartate aminotransferase level | 3, 7, 14 and 28 days
  Compare the change in aspartate aminotransferase level at 3, 7, 14 and 28 days after treatment
Change in alanin aminotransferase level | 3, 7, 14 and 28 days
  Compare the change in Alanine aminotransferase levels at 3, 7, 14 and 28 days after treatment
Change in bilirubin level | 3, 7, 14 and 28 days
  Compare the change in bilirubin levels at 3, 7, 14 and 28 days after treatment
Change in lactate dehydrogenase level | 3, 7, 14 and 28 days
  Compare the change in lactate dehydrogenase levels at 3, 7, 14 and 28 days after treatment
Change in creatine kinase level | 3, 7, 14 and 28 days
  Compare the change in creatine kinase levels at 3, 7, 14 and 28 days after treatment
Change in creatine kinase MB level | 3, 7, 14 and 28 days
  Compare the change in creatine kinase MB levels at 3, 7, 14 and 28 days after treatment
Change in C reactive protein concentration | 3, 7, 14 and 28 days
  Compare the change in C reactive protein concentration at 3, 7, 14 and 28 days after treatment, in mg/L
Change in D Dimer concentration | 3, 7, 14 and 28 days
  Compare the change in D Dimer concentration at 3, 7, 14 and 28 days after treatment
Change in Procalcitonin concentration | 3, 7, 14 and 28 days
  Compare the change in procalcitonin concentration at 3, 7, 14 and 28 days after treatment
Change in IL6 level | 3, 7, 14 and 28 days
  Compare the change in IL6 level at 3, 7, 14 and 28 days after treatment
Radiography imaging | Over a period of 60 days
  Resolution of chest radiography imaging findings (example, bilateral, peripheral and basal predominant ground-glass opacity, consolidation, or both)
Tomography imaging | Over a period of 60 days
  Resolution of tomography imaging (example, patches located in the subpleural regions of the lung)
Assessment of oxygenation | 3, 7, 14 and 28 days
  Arterial oxygen partial pressure (PaO2) in mmHg / Inspired fraction of oxygen (FIO2) ratio
Viral Load | 0, 3, 7 days and until hospital discharge or a maximum of 60 days whichever comes first
  Viral Load Quantification
Antibody titer | Day 0, Day 3 and Day 7
  Neutralizing antibody anti SARS-CoV-2 titer evolution
Oxygen-free days through Day 60 | Until hospital discharge or a maximum of 60 days whichever comes first
  Number of days without use of Oxygen
Mechanical ventilation-free days through Day 28 | Until hospital discharge or a maximum of 28 days whichever comes first
  Number of days without use of mechanical ventilation
Intensive Care Unit (ICU)-free days through Day 28 | Until hospital discharge or a maximum of 28 days whichever comes first
  Time outside of ICU, in days
Hospital-free days through Day 60 | Until hospital discharge or a maximum of 60 days whichever comes first
  Time outside of the hospital, in days

OTHER OUTCOMES:
Incidence of adverse events | Up to 28 days
  Occurrence of adverse events during inactivated convalescent plasma transfusion, classified according to the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Andrés F Zuluaga, MD, MSc, MeH, Principal Investigator — Universidad de Antioquia
Locations (10):
- Colombia (10):
  - Clínica Antioquía, Medellín, Antioquía
  - Clínica Sagrado Corazón, Medellín, Antioquía
  - IPS Universitaria, Medellín, Antioquía
  - Universidad de Antioquía, Medellín, Antioquía
  - National Blood Center Foundation, Hemolife/Fundación Banco Nacional de Sangre Hemolife, Bogotá, Cundinamarca
  - Clínica Rosales, Pereira, Risaralda Department
  - Clinica Nuestra, Cali, Valle del Cauca Department
  - Clínica Corpas, Bogotá
  - E.S.E Hospital San Rafael Facatativa, Facatativá
  - Clínica la Estancia, Popayán

REFERENCES:
- [Background] Epstein J, Burnouf T. Points to consider in the preparation and transfusion of COVID-19 convalescent plasma. Vox Sang. 2020 Aug;115(6):485-487. doi: 10.1111/vox.12939. Epub 2020 May 14. No abstract available. PMID 32319102
- [Background] Shen C, Wang Z, Zhao F, Yang Y, Li J, Yuan J, Wang F, Li D, Yang M, Xing L, Wei J, Xiao H, Yang Y, Qu J, Qing L, Chen L, Xu Z, Peng L, Li Y, Zheng H, Chen F, Huang K, Jiang Y, Liu D, Zhang Z, Liu Y, Liu L. Treatment of 5 Critically Ill Patients With COVID-19 With Convalescent Plasma. JAMA. 2020 Apr 28;323(16):1582-1589. doi: 10.1001/jama.2020.4783. PMID 32219428
- [Background] Casadevall A, Pirofski LA. The convalescent sera option for containing COVID-19. J Clin Invest. 2020 Apr 1;130(4):1545-1548. doi: 10.1172/JCI138003. No abstract available. PMID 32167489